CLINICAL TRIAL: NCT02573649
Title: Effects of Closed-loop Stimulation vs. DDD Pacing on Prevalence and Timing of Haemodynamic Variations and Clinical Prodromes Induced by Head-up Tilt Test in Patients With Refractory Cardioinhibitory Vasovagal Syncope. The TIRECS Study
Brief Title: The Tilt Test-Induced REsponse in Closed-loop Stimulation (TIRECS) Study
Acronym: TIRECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Principal Investigator, Pietro Palmisano, physician, Azienda Ospedaliera Cardinale G. Panico
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TIRECS
Record Dates: First submitted 2015-08-09; First posted 2015-10-12 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Syncope, Vasovagal, Neurally-Mediated
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLS-ON first (Active Comparator): Closed-loop Stimulation on first
  Interventions: Device: Closed-loop Stimulation on first
- CLS-OFF first (Active Comparator): Closed-loop Stimulation off first
  Interventions: Device: Closed-loop Stimulation off first

INTERVENTIONS:
Device: Closed-loop Stimulation on first — Closed-loop Stimulation algorithm is turned on in the device. The patient performs a head up tilt test. After a week Closed-loop Stimulation algorithm is turned off and the patient performs a second head up tilt test.
  Arms: CLS-ON first
Device: Closed-loop Stimulation off first — Closed-loop Stimulation algorithm is turned off in the device. The patient performs a head up tilt test. After a week Closed-loop Stimulation algorithm is turned on and the patient performs a second head up tilt test.
  Arms: CLS-OFF first

SUMMARY:
Multicentre, prospective, double blinded, randomized study designed as an intrapatient comparison to evaluate the effects of the Biotronik Closed-loop Stimulation algorithm on prevalence and timing of haemodynamic variations and clinical prodromes induced by head-up tilt test in patients underwent pacemaker implantation for refractory cardioinhibitory vasovagal syncope.

DETAILED DESCRIPTION:
A total of 30 patients with refractory cardioinhibitory vasovagal syncope receiving a Biotronik pacemaker with Closed-loop Stimulation (CLS) algorithm will be enrolled in the study. Two head-up tilt test (HUTT), one during DDD 60/min pacing with CLS algorith turned off (CLS-OFF) and the other during DDD-CLS pacing (CLS-ON), will be performed one week apart; patients will be randomly and blindly assigned to group A (n=15, first HUTT in CLS-ON mode) or B (n=15, first HUTT in CLS-OFF mode). During HUTT heart rate, blood pressure, and the incidence of clinical prodromes and syncope wil be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Refractory cardioinhibitory vasovagal syncope treated with permanent pacemaker;
* Pacemaker Biotronik with Closed-loop Stimulation algorithm
* Ability to perform a head up tilt test
* Completion of the 18th year of age

Exclusion Criteria:

* Contraindications to head up tilt test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Haemodynamic response during head up tilt test. | 45 minutes
  Assessment of the values of systolic blood pressure
Incidence of prodromal symptoms during head up tilt test. | 45 minutes
  Assessment of patient-reported symptoms during the test
Incidence of syncope during head up tilt test. | 45 minutes
  Assessment of patient-reported symptoms during the test

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Palmisano, MD, Principal Investigator — Cardiology Unit, Card G. Panico Hospital, Tricase, Italy
Locations (2):
- Italy (2):
  - Pietro Palmisano, Tricase, Lecce
  - Dell'Era Gabriele, Novara, Novara